CLINICAL TRIAL: NCT02212717
Title: Endosonography-guided Gallbladder Drainage (EGBD) Versus Percutaneous Cholecystostomy (PC) in Patients Suffering From Acute Cholecystitis That Are Unsuitable for Surgery. A Randomized Controlled Trial.
Brief Title: A Randomized Controlled Trial on EGBD vs PC for Acute Cholecystitis.
Acronym: DRAC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); Tokyo Medical University (Other); Kinki University (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC-2014.301-T
Record Dates: First submitted 2014-08-05; First posted 2014-08-08 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Acute Cholecystitis
Keywords: Acute cholecystitis; EUS-guided gallbladder drainage; Percutaneous cholecystostomy
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-guided gallbladder drainage (Active Comparator)
  Interventions: Procedure: EUS-guided gallbladder drainage (EGBD)
- Percutaneous cholecystomy (Active Comparator)
  Interventions: Procedure: Percutaneous cholecystostomy (PC)

INTERVENTIONS:
Procedure: EUS-guided gallbladder drainage (EGBD) — The gallbladder would be identified by a linear echoendoscope (EUS) and a suitable puncture site in the stomach or the duodenum without intervening blood vessels would be located. The gallbladder would be punctured with a 19-gauge needle and a guidewire would be passed through the needle and looped in the gallbladder. The Hot AXIOS stent would then be inserted. A naso-gallbladder drain or a 5-7Fr double pigtail stents can be inserted into gallbladder if the effluent failed to clear after irrigation. This would be performed to improve drainage and avoid obstruction of the stent.
  Arms: EUS-guided gallbladder drainage
Procedure: Percutaneous cholecystostomy (PC) — Trained interventional radiologists in the respective hospitals would perform the procedure under local anesthesia. A transhepatic route would be used in all patients to decrease bile leakage. An 8.5 Fr pigtail drainage catheter would be placed between the 8th or 9th intercostal space under sonographic and fluoroscopic guidance. The pigtail catheter would be drained to a bedside bag.
  Arms: Percutaneous cholecystomy

SUMMARY:
Acute cholecystitis commonly occurs in elderly patients that are high-risk candidates for surgery. Percutaneous cholecystostomy (PC) is frequently employed for gallbladder drainage in these patients. Recently, the feasibility of EUS-guided gallbladder drainage (EGBD) in treatment of this condition has been demonstrated but how the two procedures compare to one another is uncertain.

The aim of this study is to compare EGBD versus PC as a definitive treatment, in high-risk patients suffering from acute cholecystitis in a randomized controlled trial. We hypothesize that EGBD can reduce the morbidity, re-intervention and mortality when compared to PC.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged ≥ 18 years old admitted for acute cholecystitis but are unsuitable for early laparoscopic cholecystectomy due to poor premorbid conditions including: American society of anesthesiology grading ≥ 3, APACHE score ≥ 12, limited life expectancy (less than 2 years) or deemed unsuitable for general anesthesia would be included.
* Written informed consent from patient or guardian who is able to understand the nature and possible consequences of the study

Exclusion Criteria:

* Pregnancy
* Patients unwilling to undergo follow-up assessments
* Patients with suspected gangrene or perforation of the gallbladder
* Patients diagnosed with concomitant liver abscess or pancreatitis (defined as elevated serum amylase more than three times the upper limit of normal)
* Altered anatomy of the upper gastrointestinal tract due to surgery of the esophagus, stomach and duodenum
* Patients with liver cirrhosis, portal hypertension and/or gastric varices
* Abnormal coagulation: INR > 1.5 and/or platelets < 50.000/mm3
* Previous drainage of the gallbladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Overall morbidities | 1 years

SECONDARY OUTCOMES:
Technical success | 30 days
  Technical success is defined as the ability to access and drain the gallbladder by placement of a drainage tube or stent.
Pain scores | 7 days
  Pain assessment would be performed using the visual-analogue scale (1 to 100) on post-procedural days 1 to 7.
Analgesic requirements | 7 days
  The amount of analgesic consumed during admission will be recorded and compared between groups. Oral panadol and intravenous tramadol (or equivalent) would be provided as required to patients.
Stone clearance rates | 1 years
  The presence or absence of gallstones after 1 years would be assessed by abdominal ultrasonography
Clinical success | 30 days
  Clinical success is obtained when the patient is afebrile and had more than 20% decrease in white cell counts.
Reintervention rate | 1 year
  The number of patients requiring biliary related re-interventions within 1 year
Re-admission rate | 1 year
  The number of patients requiring hospital re-admissions due to biliary related events

CONTACTS AND LOCATIONS:
Locations (4):
- Chinese University of Hong Kong, Hong Kong, Hong Kong, China
- Japan (2):
  - Kinki University Hospital, Osaka
  - Tokyo Medical University Hospital, Tokyo
- University Hospital Rio Hortega, Barcelona, Spain

REFERENCES:
- [Background] de la Serna-Higuera C, Perez-Miranda M, Gil-Simon P, Ruiz-Zorrilla R, Diez-Redondo P, Alcaide N, Sancho-del Val L, Nunez-Rodriguez H. EUS-guided transenteric gallbladder drainage with a new fistula-forming, lumen-apposing metal stent. Gastrointest Endosc. 2013 Feb;77(2):303-8. doi: 10.1016/j.gie.2012.09.021. Epub 2012 Dec 1. No abstract available. PMID 23206813
- [Background] Itoi T, Binmoeller KF, Shah J, Sofuni A, Itokawa F, Kurihara T, Tsuchiya T, Ishii K, Tsuji S, Ikeuchi N, Moriyasu F. Clinical evaluation of a novel lumen-apposing metal stent for endosonography-guided pancreatic pseudocyst and gallbladder drainage (with videos). Gastrointest Endosc. 2012 Apr;75(4):870-6. doi: 10.1016/j.gie.2011.10.020. Epub 2012 Jan 31. PMID 22301347
- [Background] Teoh AY, Binmoeller KF, Lau JY. Single-step EUS-guided puncture and delivery of a lumen-apposing stent for gallbladder drainage using a novel cautery-tipped stent delivery system. Gastrointest Endosc. 2014 Dec;80(6):1171. doi: 10.1016/j.gie.2014.03.038. Epub 2014 May 13. No abstract available. PMID 24830582
- [Derived] Teoh AYB, Kitano M, Itoi T, Perez-Miranda M, Ogura T, Chan SM, Serna-Higuera C, Omoto S, Torres-Yuste R, Tsuichiya T, Wong KT, Leung CH, Chiu PWY, Ng EKW, Lau JYW. Endosonography-guided gallbladder drainage versus percutaneous cholecystostomy in very high-risk surgical patients with acute cholecystitis: an international randomised multicentre controlled superiority trial (DRAC 1). Gut. 2020 Jun;69(6):1085-1091. doi: 10.1136/gutjnl-2019-319996. Epub 2020 Mar 12. PMID 32165407